CLINICAL TRIAL: NCT01092741
Title: Therapy of Late Chronic Phase Chronic Myelogenous Leukemia (CML) With High-Dose Gleevec (STI571)
Brief Title: Late Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-292
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: Leukemia; Gleevec; STI571; CML; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gleevec (Experimental): Gleevec 400 mg by mouth (P.O.) twice daily = 800 mg total daily dose
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — 400 mg P.O. twice daily (800 mg total daily dose)
  Other Names: STI571

SUMMARY:
Objectives:

Primary endpoints:

To achieve low levels of Polymerase Chain Reaction (PCR) ratios of B-cell antigen receptor (Bcr-Abl)/Bcr (molecular CR) in a significant proportion of patients after 12 months of higher doses (800 mg daily) of Gleevec therapy To increase the proportion of patients achieving a complete cytogenetic response in patients with Ph-positive chronic phase CML using initial higher dose Gleevec therapy.

Secondary endpoints:

To evaluate the durations of PCR negativity, cytogenetic response, hematologic control, and survival.

To analyze differences in response rates and in prognosis within different risk groups and patient characteristics

DETAILED DESCRIPTION:
Treatment: Imatinib mesylate is a new oral medication that blocks a protein that is responsible for CML

Patients on this study will take 400 mg of imatinib twice daily (morning and evening). If you have side effects, the dose may be lowered. If you are taking less than 800 mg of imatinib, you can take your dose once per day or divided in two doses. Imatinib mesylate should be taken with a large glass of water.

After completing 3 to 12 months of therapy, response to imatinib mesylate will be evaluated. Treatment may be continued for up to 20 years, or as long as it is judged best to control the leukemia.

Update June 2010:

Blood tests are recommended 2 times per year. Your doctor will discuss with you how often you should have blood tests. Bone marrow will be done if your doctor thinks it is necessary to check your disease. You must return to M. D. Anderson at least once every year. You may not need a bone marrow test every visit, but you will have blood drawn to measure the amount of disease you have. If the leukemia cannot be found for 2 years or longer on the blood test called PCR which is done to measure the amount of disease you have, your doctor may talk to you about stopping treatment with imatinib. If you and your doctor decide to stop your therapy, you will have a blood test for PCR done every 3 to 6 months. You do not need to return to M. D. Anderson to have this blood test done. You may have the blood taken by your local doctor and mailed to M. D. Anderson. If the leukemia is found again by the PCR blood test, your doctor may recommend that you restart treatment with imatinib. You may decide to stay on treatment with imatinib even if your PCR blood test does not show any sign of leukemia for 2 years or longer.

This is an investigational study. The FDA has authorized the use of imatinib mesylate for patients with CML. It is the dose of imatinib mesylate being used that is investigational. A total of 50 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 15 years or older with a diagnosis of Ph-positive or Bcr-positive CML in chronic phase CML. They should be in at least one of the categories below: A. Patients must have received interferon alpha and: - Failed to achieve or lost a hematologic complete remission(after 3 months of therapy with interferon), or - Failed to achieve or lost a major cytogenetic remission, or - Failed to achieve or lost a complete molecular remission (competitive quantitative PCR <0.05%), or - Were intolerant to interferon B. Patients in late chronic phase (i.e., >/= 12 months from diagnosis) who have not received treatment with interferon and: - Have high risk for toxicity with IFN-A (e.g., age >/= 60 years), or - Refuse to use IFN-A
2. ECOG performance of 0-2.
3. Serum bilirubin less than 2mg%, serum creatinine less than 2mg%.

Exclusion Criteria:

1. - NYHA Class 3-4 heart disease; Pregnant or lactating females
2. Women of pregnancy potential must practice contraception
3. Patients in accelerated phase (except clonal evolution) or blastic phase are excluded. - Patients with clonal evolution as their only criterion for accelerated phase are eligible.
4. Inclusion of women and minorities: As per NIH policy, women and members of minorities will be included in this protocol as they are referred in the CML population.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2001-07; Primary Completion 2006-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cytogenetic Complete Response (CR) Rate | Evaluated at 6 months; Polymerase Chain Reaction (PCR) testing for BCR-ABL every 3-4 months in year one then every year.
  CR Rate = Number participants out of total treated with complete cytogenetic response. Complete Hematologic Remission (CHR) - normalization >4 weeks of bone marrow (less than 5% blasts) & peripheral blood with white blood count (WBC)<10x10^9/L & no peripheral blasts, promyelocytes or myelocytes, disappearance of all signs & symptoms of disease. Partial Hematologic Response (PHR) = CHR except persistence of immature cells (myelocytes, metamyelocytes), or splenomegaly <50% of pretreatment, or thrombocytosis >450x10^9/L but <50% of pretreatment. Complete hematologic remission further classified according to suppression of Philadelphia chromosome (Ph) by cytogenetics or fluorescence in situ hybridization (FISH): a) No cytogenetic response - Ph positive 100% of pretreatment value; b) Minor cytogenetic response - Ph positive 35-90% of pretreatment value; c) Partial cytogenetic response - Ph positive 1-34% of pretreatment value; d) Complete cytogenetic response - Ph positive 0%.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — The University Of MD Anderson Cancer Center
Locations (1):
- The University Of MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center web site — http://www.mdanderson.org